CLINICAL TRIAL: NCT02339844
Title: Pan European Collaboration on Antipsychotic Naïve Schizophrenia II
Acronym: PECANSII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Birte Glenthoj, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2013-149
Record Dates: First submitted 2014-12-08; First posted 2015-01-16 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia
Keywords: glutamate; dopamine; cognition; cortical thickness; ppi; p50
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antipsychotic treatment (Active Comparator): individual doses of aripiprazole for all patients
  Interventions: Drug: Aripiprazole
- no treatment (No Intervention): no treatment for all healthy controls

INTERVENTIONS:
Drug: Aripiprazole — 6 weeks of individual doses of aripiprazole
  Other Names: Abilify
  Arms: antipsychotic treatment

SUMMARY:
The study is a prospective 2 year multimodal follow-up study of initially antipsychotic-naïve first-episode psychotic patients involving a standardized intervention with monotherapy with aripiprazole during the first 6 weeks. Patients and matched healthy controls will be examined after 6 weeks, 6 months and 2 years. They will be examined with MR-scannings, neurocognitive tests, EEG, and PET-scannings.

DETAILED DESCRIPTION:
The study is a prospective 2 year multimodal follow-up study of initially antipsychotic-naïve first-episode psychotic patients involving a standardized intervention with monotherapy with aripiprazole during the first 6 weeks. Patients and matched healthy controls will be examined at baseline and after 6 weeks, 6 months and 2 years.

Levels of glutamate and gamma-aminobutyric acid (GABA) are measured by proton magnetic resonance spectroscopy (1H-MRS) in the anterior cingulate cortex ACC and thalamus. Presynaptic Dopamine level is measured with Positron Emission Tomography Computed Tomography (PET/CT)-scanning using 3,4-dihydroxy-6-[18F]fluoro-L-phenylalanine (18F-DOPA). Disturbances of the reward system is measured with functional magnetic resonance imaging (fMRI) . Regional cerebral blood flow and activity in the same regions are measured with Pseudo-continuous arterial spin labelling (pCASL). The default mode network, functional and structural connectivity in the associated macro circuits are measured with resting state fMRI, EEG, and diffusion tensor imaging. Structural brain changes (in grey and white matter) are measured with MRI. Cognitive functions are measured with a neuropsychological test battery, and early information processing with event related EEG and electromyography (EMG) (psychophysiological examinations). Further patients psychopathology will be rated.

ELIGIBILITY:
Inclusion Criteria Patients:

* Fulfilling the diagnostic criteria of schizophrenia or schizoaffective disorder according to ICD-10 (International Classification of Diseases version 10) or DSM-IV/V (Diagnostic and Statistical Manual version 4 /5)
* Age 18-45 years
* Never treated with antipsychotic compounds or central nervous system (CNS) stimulants
* Legally competent

Inclusion criteria controls:

* Matching patients on age (+/- 2 years), sex and parental socioeconomic status
* Age 18-45 years
* No psychiatric or physical disease

Exclusion Criteria patients:

* Substance abuse on a daily basis during the last 3 month or patients fulfilling the criteria of ongoing substance abuse due to ICD-10/DSM-IV/V
* Treatment with antidepressant during the last 30 days
* Head injury with more than 5 minutes of unconsciousness
* Patients involuntarily admitted or treated
* Components of metal implanted by operation
* Pacemaker
* Pregnancy
* Severe physical illness

Exclusion criteria controls

* First degree relatives with psychiatric disease
* Substance abuse during the last 3 month or positive screening of drugs in urine-sample
* Head injury with more than 5 minutes of unconsciousness
* Components of metal implanted by operation
* Pacemaker
* Pregnancy
* Severe physical illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2014-01; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Glutamate level in Anterior Cingulate Cortex (measured with magnetic resonance spectroscopy) | Baseline, 6 weeks, 6 months, 2 years
  Glutamate level at baseline and change over time as measured with magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Cortical thickness (measured with magnetic resonance and free surfer) | Baseline, 6 weeks, 6 months & 2 years
  Thickness of grey matter measured with magnetic resonance and free surfer
Dopamine syntheses capacity in striatum (measured with F-DOPA using Positron emission tomography) | Baseline and 6 weeks follow up
  Dopamine measured with F-DOPA using Positron emission tomography
Reward system activation in striatum (measured with functional magnetic resonance imaging) | Baseline and 6 weeks follow up
  Reward activity is measured with functional magnetic resonance imaging
Neurocognition (measured with BACS (Brief Assessment of Cognition in Schizophrenia) and CANTAB (Cambridge Neuropsychological Test Automated Battery) | Baseline, 6 weeks, 6 months & 2 years
  Neurocognition is measured with BACS (Brief Assessment of Cognition in Schizophrenia) and CANTAB (Cambridge Neuropsychological Test Automated Battery)
Psychopathology (measured with PANSS (Positive and Negative Syndrome Scale) | Baseline, 6 weeks, 6 months & 2 years
  Psychopathology is measured with PANSS (Positive and Negative Syndrome Scale)
Prepulse inhibition of the startle reflex and reduced P50 suppression ( measured with event related EEG and EMG) | Baseline, 6 weeks, 6 months & 2 years
  Disturbances in early information processing in form of impaired sensory filtering as measured with event related EEG and EMG

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthøj, Professor, Study Director — Capital Mental Health Services, Center for Neuropsykiatrisk Skizofreniforskning, CNSR & Lundbeck Foundation Center for Clinical Intervention and Neuropsychiatric Schizophrenia Research, CINS
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Centre Glostrup, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bojesen KB, Ambrosen KS, Sigvard AK, Nielsen MO, Gjedde A, Kumakura Y, Jensen LT, Fuglo D, Ebdrup BH, Rostrup E, Glenthoj BY. Interrelations between dopaminergic-, gabaergic- and glutamatergic neurotransmitters in antipsychotic-naive psychosis patients and the association to initial treatment response. Mol Psychiatry. 2025 Sep 12. doi: 10.1038/s41380-025-03229-0. Online ahead of print. PMID 40940558
- [Derived] Bojesen KB, Broberg BV, Fagerlund B, Jessen K, Thomas MB, Sigvard A, Tangmose K, Nielsen MO, Andersen GS, Larsson HBW, Edden RAE, Rostrup E, Glenthoj BY. Associations Between Cognitive Function and Levels of Glutamatergic Metabolites and Gamma-Aminobutyric Acid in Antipsychotic-Naive Patients With Schizophrenia or Psychosis. Biol Psychiatry. 2021 Feb 1;89(3):278-287. doi: 10.1016/j.biopsych.2020.06.027. Epub 2020 Jul 10. PMID 32928500
- [Derived] Jessen K, Mandl RCW, Fagerlund B, Bojesen KB, Raghava JM, Obaid HG, Jensen MB, Johansen LB, Nielsen MO, Pantelis C, Rostrup E, Glenthoj BY, Ebdrup BH. Patterns of Cortical Structures and Cognition in Antipsychotic-Naive Patients With First-Episode Schizophrenia: A Partial Least Squares Correlation Analysis. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 May;4(5):444-453. doi: 10.1016/j.bpsc.2018.09.006. Epub 2018 Sep 25. PMID 30420252
- See also: additional information — https://www.psykiatri-regionh.dk/cinsr/Pages/default.aspx